CLINICAL TRIAL: NCT04598594
Title: Evaluation of the Efficacy of Nicotine Patches in SARS-CoV2 (COVID-19) Infection in Intensive Care Unit Patients
Acronym: NICOVID-REA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200537; 2020-003723-42 (EudraCT Number)
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Covid19; SARS-Associated Coronavirus as Cause of Disease Classified Elsewhere
Keywords: Covid19; SARS-CoV2; Mechanical ventilation; ICU; Nicotine
MeSH Terms: conditions — COVID-19 | interventions — Tobacco Use Cessation Devices; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine patch (Experimental)
  Interventions: Drug: Patch, Nicotine
- Placebo patch (Placebo Comparator)
  Interventions: Drug: Patch, Placebo

INTERVENTIONS:
Drug: Patch, Nicotine — Two patches of 7 mg/day Treatment at 14 mg/day during mechanical ventilation since after first successful extubation then, dose decreasing: Week 1: 10,5 mg/day Week 2 : 7 mg/day Week 3 : 3,5 mg/day
  Arms: Nicotine patch
Drug: Patch, Placebo — Two patches of 7 mg/day Treatment at 14 mg/day during mechanical ventilation since after first successful extubation then, dose decreasing: Week 1: 10,5 mg/day Week 2 : 7 mg/day Week 3 : 3,5 mg/day
  Arms: Placebo patch

SUMMARY:
There is currently no known treatment for COVID19. Active smokers are infrequent among patients with COVID-19 which has led our team to hypothesize that nicotine is responsible for this protective effect via the nicotinic acetylcholine receptor (nAChR). In fact, nAChR possess the ability to modulate ACE2 expression, the cellular doorway for SARS-CoV2. nAChR modulation by the virus would be responsible for the numerous clinical signs observed in COVID-19, including the cytokine storm manifested in intensive care hyperinflammatory patients.

Based on epidemiological data and experimental data from scientific literature, our team hypothesize that nicotine could inhibit the penetration and propagation of SARS-CoV2. Our team also claim that nicotine could attenuate the hyperinflammatory response and cytokine storm leading to acute respiratory failure and a probable multi-organ failure associated with COVID19.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years
2. Documented diagnosis of COVID 19 (according to the tests referenced on the list published on the website : https://covid-19.sante.gouv.fr.tests)
3. Hospitalized in intensive care unit, intubated and mechanically ventilated for less than 48 hours
4. Non-smoker and non-vaping or abstinent patient for at least 12 months
5. Obtain written informed consent from a relative / relative / support person. In the absence of a close/relative/trusted person, the patient may be included according to the emergency procedure by the investigating doctor.
6. Affiliated to a social security scheme or beneficiary of such a scheme (AME excluded)

Exclusion Criteria:

1. Chronic respiratory failure defined by PaCO2> 60 mmHg in ambulatory patients (respiratory parameters at baseline).
2. Mechanical ventilation at home (non-invasive mechanical ventilation or via a tracheostomy) with the exception of CPAP / BIPAP used only for sleep apnea syndromes
3. Predictable mechanical ventilation duration <48 hours
4. Moribund patient or death expected on the day of randomization, or with a SAPS II score> 90
5. Cerebral deficiency with dilated areactive pupils or irreversible neurological pathology.
6. Other concomitant severe pathology with an estimated life expectancy of less than 1 year
7. Treatment with nicotine replacement therapy or varenicline or bupropion ongoing
8. Contraindication for nicotine patches:

   * Pregnant or breastfeeding women
   * Allergy to nicotine or to one of the excipients of the transdermal patch
   * Generalized skin pathologies
   * Cerebrovascular accident or acute coronary syndrome for less than 3 months
   * Pheochromocytoma
   * Unstable or worsening angor
   * Severe cardiac arrhythmia (Defined by wearing an automatic implantable defibrillator)
   * Known severe heart failure (Defined, for this study, by systolic LV dysfunction with an LV ejection fraction (LVEF) of less than 30%)
   * Severe renal failure (Defined by KDIGO stage 3)
   * Severe hepatic impairment (Defined by a factor V <30%)
   * Arteriopathy obliterating of the lower limbs stage III and IV
   * Uncontrolled hyperthyroidism
   * Gastroduodenal esophagitis or ulcer undergoing treatment or active
9. Patient under guardianship or curatorship
10. Patient deprived of liberty by judicial or administrative decision
11. Patient included in another interventional trial evaluating a health product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 28

SECONDARY OUTCOMES:
Mortality | Day 60
Time before successful extubation | Day 60
  Without reintubation or death in the following 48 hours for tracheotomized patients: alive and not ventilated for 48 hours (with death and LATA in competitive risks).
Number of days living without invasive mechanical ventilation | Day 28
Composite score incorporating death and the number of days living without mechanical ventilation | Day 60
  This is a ranked composite score that incorporates death and days free from mechanical ventilation through day 28, calculated in such a manner that death constitutes a worse outcome than fewer days off the ventilator.16 Time free from mechanical ventilation was calculated as the number of days between successful liberation from the ventilator and study day 60. Each patient was compared with every other patient in the study and assigned a score (tie: 0, win: +1, loss: -1) for each pairwise comparison based on whom fared better
Mean evolution of blood gases | Day 1 to Day 14
  measured each day from day 1 to day 14
Mean evolution of Tidal Volume (ventilator parameters) | Day 1 to Day 14
  measured each day from day 1 to day 14
Mean evolution of respiratory rate (ventilator parameters) | Day 1 to Day 14
  measured each day from day 1 to day 14
Mean evolution of Positive Expiratory Pressure (ventilator parameters) | Day 1 to Day 14
  measured each day from day 1 to day 14
Mean evolution of plateau pressure (ventilator parameters) | Day 1 to Day 14
  measured each day from day 1 to day 14
Mean evolution of fraction of inspired oxygen (ventilator parameters) | Day 1 to Day 14
  measured each day from day 1 to day 14
Evolution of the Sequential Organ Failure Assessment (SOFA) score and its components by organ | Day 1 to Day 28
  A higher score indicate a worse outcome
Number of days alive without organ failure | Day 28, day 60
Duration of hospitalization in intensive care unit | From day 1 up to 3 months
Duration of hospitalization in hospital | From day 1 up to 3 months
Number of days alive and out of the ICU and hospital | Day 28, day 60
Evolution of viral load | Day 7, Day 14 or day of ICU discharge if before day 14
  samples taken on D7 and D14 or the day of discharge from intensive care unit if before D14
Proportion of active smoker or active vapers or taking nicotine substitutes documented by examination | 2 weeks after treatment decrease, 8 weeks after treatment decrease
Proportion of active smoker or active vapers or taking nicotine substitutes documented by urinary cotinine | 2 weeks after treatment decrease, 8 weeks after treatment decrease
Mean score of Desire to smoke defined by French Tobacco Craving scale | 2 weeks after treatment decrease, 8 weeks after treatment decrease
Mean score of Withdrawal symptoms scale | 2 weeks after treatment decrease, 8 weeks after treatment decrease
Mean score of Hospital anxiety and depression scale | 2 weeks after treatment decrease, 8 weeks after treatment decrease
Post traumatic stress disorder scale | 2 weeks after treatment decrease, 8 weeks after treatment decrease
Mean score of Insomnia severity scale | 2 weeks after treatment decrease
Cotinin rate in blood | 8 weeks after treatment decrease

CONTACTS AND LOCATIONS:
Overall Officials: Alain COMBES, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (18):
- France (18):
  - Centre Hospitalier Victor Dupouy - Service de Réanimation polyvalente et USC, Argenteuil
  - CHRU de Besançon - Service de Médecine Intensive Réanimation, Besançon
  - Centre Hospitalier Sud Francilien - Service de réanimation, Corbeil-Essonnes
  - CHU Dijon - Hôpital François Miterrand Service de Médecine Intensive Réanimation, Dijon
  - Hôpital Simone VEIL - Service d'Anesthésie-Réanimation, Eaubonne
  - Grand Hôpital de l'Est Francilien - Site Jossigny - Réanimation, Jossigny
  - Hôpital Bicêtre - Service de Médecine Intensive Réanimation, Le Kremlin-Bicêtre
  - Grand Hôpital de l'Est Francilien Site Meaux - Service de Réanimation Médico-Chirurgicale, Meaux
  - Groupement Hospitalier de la Région de Mulhouse Sud Alsace - Hop Emile MULLER, Mulhouse
  - CHU Nice - Hôpital L'Archet 1 - Service de Médecine Intensive Réanimation, Nice
  - CHR Orléans Service de Médecine Intensive Réanimation, Orléans
  - Hôpital Pitié Salpêtrière - ICU, Paris
  - Hôpital Pitié Salpêtrière - Intensive care unit, Paris
  - Institut Mutualiste Montsouris Service de Réanimation Polyvalente, Paris
  - Hôpital Tenon - Service de Médecine Intensive Réanimation, Paris
  - Centre Hospitalier René Dubos - Service de Réanimation Médico-Chirurgicale, Pontoise
  - Hôpital DELAFONTAINE Service de Médecine Intensive Réanimation, Saint-Denis
  - Médipôle Hôpital Privé - MHP Service de Médecine Intensive Réanimation, Villeurbanne

REFERENCES:
- [Derived] Labro G, Tubach F, Belin L, Dubost JL, Osman D, Muller G, Quenot JP, Da Silva D, Zarka J, Turpin M, Mayaux J, Lamer C, Doyen D, Chevrel G, Plantefeve G, Demeret S, Piton G, Manzon C, Ochin E, Gaillard R, Dautzenberg B, Baldacini M, Lebbah S, Miyara M, Pineton de Chambrun M, Amoura Z, Combes A; NICOVID-REA Trial Group. Nicotine patches in patients on mechanical ventilation for severe COVID-19: a randomized, double-blind, placebo-controlled, multicentre trial. Intensive Care Med. 2022 Jul;48(7):876-887. doi: 10.1007/s00134-022-06721-1. Epub 2022 Jun 9. PMID 35676335